CLINICAL TRIAL: NCT04186208
Title: Prospective, Non-interventional Study to Evaluate the Efficacy and Safety of NOVOCART® 3D for the Treatment of Cartilage Defects of the Knee in Pediatric Patients With Closed Epiphyses
Brief Title: Non-interventional Study With NOVOCART® 3D for the Treatment of Cartilage Defects of the Knee in Pediatric Patients
Acronym: JUNOVO
Status: Active, not recruiting | Type: Observational
Sponsor: Tetec AG (Industry)
Collaborators: Aesculap AG (Industry); Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1633
Record Dates: First submitted 2019-01-07; First posted 2019-12-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cartilage Disease
Keywords: cartilage defect; knee; pediatric patients
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: NOVOCART 3D — Autologous Chondrocyte Implantation

SUMMARY:
Prospective, multicenter, single-arm non-interventional study to evaluate the efficacy, safety and health economics of NOVOCART 3D in the Treatment fo cartilage defects of the knee in pediatric patients wieh closed epiphyseal growth plates.

DETAILED DESCRIPTION:
The present study is a prospective, multicenter, single-arm non-interventional study to evaluate the efficacy, safety and health economics of NOVOCART® 3D in the treatment of cartilage defects of the knee in pediatric patients with closed epiphyseal growth plates.

In this non-interventional study NOVOCART® 3D, which is marketed in Germany under Paragraph 4b Medicinal Products Act, will be used in routine clinical practice according to the authorized Summary of Product Characteristics (SmPC). As stated in this SmPC, NOVOCART® 3D may only be used by physicians who are trained on the product. The treatment with NOVOCART® 3D requires two surgeries. During the first surgery cartilage biopsies will be harvested arthroscopically and sent to TETEC AG (Tissue Engineering Technologies AG) for NOVOCART® 3D manufacturing, then NOVOCART® 3D will be transplanted during a second surgery about 3 to 4 weeks later.

All patients will be followed up for 5 years post NOVOCART® 3D transplantation and data will be collected at 3, 6, 12, 18, 24, 36, 48 and 60 months as outlined at the end of this synopsis.

NOVOCART® 3D post treatment rehabilitation should follow the recommendations given in the SmPC and during product training.

The primary and secondary variables (see below) will be assessed after a follow-up of 24 month post NOVOCART® 3D transplantation (primary analysis).

Long-term data will be assessed after an additional 3 years follow-up (follow-up analysis).

The collected data will be documented using dedicated case report forms (CRFs) which are created and printed by TETEC AG.

ELIGIBILITY:
Inclusion Criteria:

* 13 - 17 years old
* Medicinal indication for NOVOCART 3D treatment

Exclusion criteria:

• none

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will include pediatric patients (< 18 years of age) with closed epiphyses who suffer from a full-thickness cartilage defect of the knee caused by acute or repetitive trauma or by osteochondritis dissecans and who are scheduled for treatment with NOVOCART® 3D. Further inclusion/exclusion criteria are given in the current version of the NOVOCART® 3D SmPC, where the therapeutic indications, contraindications, special warnings and precautions for use are listed in detail.
  The decision to treat patients with NOVOCART® 3D must be made independently from the patient's participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of Overall KOOS (Knee Injury and Osteoarthritis Outcome Score) | 24 months Follow Up (FU)
  Change of KOOS defined as the average of the 5 subscale scores (range 0-100, higher values represent a better outcome)

SECONDARY OUTCOMES:
Change of 5 subscores KOOS | 24 months FU
  Change of the 5 subscores of KOOS (range 0-100, higher values represent a better outcome)
IKDC subjective | 24 month FU
  Change of IKDC (International Knee Documentation Committee) subjective (range 0-100, higher values represent a better outcome)
pain VAS | 24 month FU
  Change in pain VAS (Visual Analogue Scale) (range 0-10, higher values represent a better outcome)
MOCART | 24 month FU
  In vivo Performance via MRI (Magnetic Resonance Imaging), MOCART Score (Magnetic Resonance Observation of Cartilage Repair Tissue) (range 0-100, higher values represent a better outcome)
KOOS responder rate | 24 month FU
  KOOS responder rate defined as Proportion of patients with > 10 Points improvement in KOOS
IKDC subjective responder rate | 24 months FU
  IKDC subjective responder rate defined as Proportion of patients with >20.5 Points improvement in IKDC subjective
Proportion of patients with Treatment failures | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Proportion of patients with Treatment failures
Health economics variable (Days of missing work/school ) to NOVOCART 3D treatment | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Days of missing work/school due to knee pain/function issues in the target knee
Health economics variable (Days of hospitalization ) to NOVOCART 3D treatment | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Days of hospitalization due to knee pain/function issues in the target knee
Health economics variable (Number of postoperative doctor visits) to NOVOCART 3D treatment | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Number of postoperative doctor visits

CONTACTS AND LOCATIONS:
Overall Officials: Peter Angele, Prof. MD, Principal Investigator — Universitätsklinikum Regensburg
Locations (6):
- Germany (6):
  - Theresienkrankenhaus und St. Hedwig-Klinik GmbH, Mannheim, Baden-Wurttemberg
  - Sportklinik Stuttgart, Stuttgart, Baden-Wurttemberg
  - Klinik und Poliklinik für Orthophädie, Physikalische Medizin und Rehabilitation Knie- und Schulterorthopädie, München, Bavaria
  - Klinikum rechts der Isar der technischen Universität München, München, Bavaria
  - Univerisätsklinikum Regensburg, Regensburg, Bavaria
  - Lubinus Clinicum Kiel, Kiel, Schleswig-Holstein